CLINICAL TRIAL: NCT06714461
Title: Post Authorization Safety Study on Assessment of Effectiveness of Additional Risk Minimization Measures Related to ARAVA® (Leflunomide) in Saudi Arabia
Brief Title: A Study of the Effectiveness of Additional Risk Minimization Measures Related to ARAVA® (Leflunomide) in Saudi Arabia
Acronym: ARAVA PASS
Status: Active, not recruiting | Type: Observational
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: OBS18508; U1111-1311-1317 (Registry Identifier: WHO ICTRP)
Record Dates: First submitted 2024-11-27; First posted 2024-12-03 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Rheumatoid Arthritis; Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis, Psoriatic | interventions — Leflunomide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Leflunomide: Participants are healthcare professionals in Saudi Arabia completing a survey regarding experience prescribing/managing/dispensing leflunomide
  Interventions: Drug: Leflunomide

INTERVENTIONS:
Drug: Leflunomide — This study will not administer any treatment, only observe the treatment as prescribed in real-world clinical practices.
  Other Names: ARAVA®

SUMMARY:
The main objective of this post-authorization safety study is to assess healthcare professionals' awareness, knowledge, and behavior related to receipt and reading of the Direct Healthcare Professional Communication and educational materials for ARAVA® (leflunomide) and of the additional risk minimization measures.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare professionals working only in Saudi Arabia
* For Prescribers: Orthopedics, Internists, Family Physicians, General Practitioners, Dermatologists, Obstetricians/Gynecologists, Immunologists, and Rheumatologists who prescribed leflunomide to women of childbearing potential in the six months preceding the time of the inclusion
* For Prescribers: Physicians or pharmacists who have prescribed or dispensed leflunomide in a pre-specified period of the 6 months leading up to survey completion
* For Pharmacists: Pharmacists (including clinical pharmacists) who have dispensed leflunomide to women of childbearing potential in the six months preceding the time of the inclusion

Exclusion Criteria:

* Healthcare professionals who may have conflicts of interest with the survey (i.e., employed by regulatory bodies or pharmaceutical companies)
* Healthcare professionals (with a relative) involved in leflunomide -related lawsuits or associations for victims of leflunomide syndrome
* Healthcare professionals who are not prescribing leflunomide
* Healthcare professionals who have prescribed or dispensed leflunomide earlier than 6 months before the survey completion

The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: In this survey-based study, the data will be collected from each healthcare professional participant in Saudi Arabia once at a certain time. However, the study will take 7 months, from 30 November 2024 to 30 May 2025, to collect the required number of responses.
Sampling Method: Non-Probability Sample
Enrollment: 3500 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2025-11-28 (Estimated); Study Completion 2025-12-03 (Estimated)

PRIMARY OUTCOMES:
Number of healthcare professionals who recall receiving and reading the additional risk minimization measures material for leflunomide distributed in 2022 | 7 months
Number of healthcare professionals aware of the information reported in the educational materials and additional risk minimization measures material distributed in 2022 | 7 months
Number of healthcare professionals reported counseling their patients and conducting the needed laboratory investigations according to 2022 additional risk minimization measures material | 7 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sanofi-Aventis, Chilly-Mazarin, France

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org